CLINICAL TRIAL: NCT05864846
Title: A Phase 4, Interventional, Multicenter, Open-Label, Single-Arm Study to Assess Behavioral and Other Co-occurring Outcomes Following Treatment With EPID(I/Y)OLEX as Add-on Therapy in Participants (Aged 1 to 65 Years Old) With Seizures Associated With Tuberous Sclerosis Complex
Brief Title: A Study to Investigate Behavioral and Other Co-Occurring Outcomes With Epidiolex as Add-On Therapy in Participants Aged 1 to 65 Years of Age With Tuberous Sclerosis Complex
Acronym: EpiCom
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JZP926-402; 2023-507426-17 (Other: EU CTR)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Tuberous Sclerosis Complex Associated Neuropsychiatric Disease
Keywords: Seizures; Tuberous Sclerosis Complex (TSC); Tuberous Sclerosis Complex Associated Neuropsychiatric Disorders (TAND); Epidiolex; Epidyolex; GWP42003-P; JZP926; TSC Associated Neuropsychiatric Disorders; Cannabidiol; Behavior
MeSH Terms: conditions — Seizures; Tuberous Sclerosis; Behavior | interventions — Cannabidiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol Oral Solution (Experimental): Participants who will receive the Cannabidiol Oral Solution (CBD-OS) titrated up to a dose of 12.5 mg/kg administered twice daily for a total dose of up to 25 mg/kg/day for 26 consecutive weeks. Participants will have the option to continue receiving the CBD-OS for an additional 26 weeks, for a total of 52 weeks.
  Interventions: Drug: Cannabidiol Oral Solution [Epidiolex]

INTERVENTIONS:
Drug: Cannabidiol Oral Solution [Epidiolex] — 100 mg/ml Cannabidiol Oral solution
  Other Names: Epidiolex

SUMMARY:
The purpose of this study is to investigate behavioral and other co-occurring outcomes with EPID(I/Y)OLEX as an add-on therapy in participants aged 1 to 65 years with tuberous sclerosis complex (TSC) who experience seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Is within the required age range at the time of signing (or at the time of the participant's parent(s)/Legally Authorized Representative (LAR) signing) the informed consent or providing assent (as applicable):

   * Participants based in the US: 1 to 65 years of age, inclusive.
   * Participants based outside the US: 2 to 65 years of age, inclusive.
2. Has a confirmed clinical diagnosis of TSC with a history of seizures in accordance with the 2012 International Tuberous Sclerosis Complex Consensus Conference criteria.
3. Has behaviors (eg, aggression, impulsivity, temper tantrum, self-injury, hyperactivity, extreme shyness, mood swings, poor eye contact, repetitive behaviors, restlessness, difficulty getting along with peers, rigid/inflexible to procedure and/or change) that are considered moderate or severe per the CareGI-S at Screening.
4. Is taking 1 or more anti-seizure medicine (ASM) at a dose that has been stable for at least 4 weeks prior to Screening.

   • All medications or interventions for epilepsy (including ketogenic diet and any neurostimulation devices for epilepsy) must have been stable for 4 weeks prior to screening and any major changes to treatment regimens should be discussed with the medical monitor.
5. Is naïve to CBD-OS treatment or has been off CBD-OS treatment for at least 3 months prior to Screening.
6. Is willing to maintain any factors expected to affect seizures stable (eg, alcohol consumption, smoking, concomitant medication usage).
7. Is male or female

   1. Male participants:

      • Male participants are eligible to participate if they agree to the following during the intervention period and for at least 2 weeks, corresponding to the time needed to eliminate the study intervention after the last dose of study intervention:
      * Refrain from donating fresh unwashed semen. PLUS
      * Use a male condom in addition to a second method of acceptable contraception used by their female partners when having sexual intercourse with a women of childbearing potential (WOCBP) who is not currently pregnant.
   2. Female participants:

      * A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

        * Is a woman of nonchildbearing potential. OR
        * Is a WOCBP and using a contraceptive method that is highly effective, preferably with low user dependency during the study intervention period and for at least 3 months after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (eg, noncompliance, recently initiated) in relationship to the first dose of study intervention.
      * A WOCBP must have a negative highly sensitive pregnancy test within 28 days before the first dose of study intervention.

Exclusion Criteria:

1. Has a clinically significant unstable medical condition other than epilepsy.
2. Has an illness during the 4 weeks prior to screening other than epilepsy which, in the investigator's opinion, could affect study outcomes.
3. Has TSC-specific tumor growth which, in the investigator's opinion, could affect the effectiveness endpoints.
4. Has previously undergone significant surgery for epilepsy that, in the investigator's opinion, may impact the assessment of outcomes.
5. Has initiated felbamate within the last 12 months prior to Screening.
6. Is currently using or has in the past used recreational or medicinal cannabis or synthetic cannabinoid-based medications within the 3 months prior to Screening and is not willing to undergo a 1-month washout period before being rescreened.
7. Has received an investigational medicinal product within the 3 months prior to the Screening Visit.
8. Has previously been assigned study intervention for this study or is currently enrolled in any other interventional study.
9. Has laboratory values at the Baseline Visit that are abnormal and of clinical significance in the investigator's opinion.
10. Participant has significantly impaired hepatic function at the Baseline Visit.
11. Has any history of suicidal behavior or any suicidal ideation of type 4 or 5 as evaluated with C-SSRS or Children's C-SSRS at the Screening Visit (for participants ≥ 4 years of age).
12. Has any known or suspected hypersensitivity to cannabinoids or any of the excipients of CBD-OS.
13. Has a known or suspected history of alcohol or substance abuse.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Change in the most problematic behavior Numerical Rating Score (NRS) score within the TAND-SQ | Baseline, Week 13, Week 26, Week 52
Change in Tuberous Sclerosis Complex Associated Neuropsychiatric Disorders Self-report, Quantified Checklist (TAND-SQ) score | Baseline, Week 13, Week 26, Week 52
Change in Aberrant Behavior Checklist (ABC) score | Baseline, Week 13, Week 26, Week 52
Change in Child Behavior Checklist (CBCL) score | Baseline, Week 26, Week 52
Change in Adult Behavior Checklist (ABCL) score | Baseline, Week 26, Week 52
Change in Adult Self-Report (ASR) score | Baseline, Week 26, Week 52
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) domains score | Baseline, Week 26, Week 52
Change in sleep characteristics using the Children's Sleep Habits Questionnaire (CSHQ) | Baseline, Week 26
Change in sleep characteristics using the Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 26
Change in executive function using Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, Week 26
Change in caregiver-reported assessment of Quality of Life (QOL) using Pediatric Quality of Life Survey Family Impact Module (PedsQL FIM) | Baseline, Week 26
Change in caregiver-reported assessment of family functioning using Pediatric Quality of Life Survey Family Impact Module (PedsQL FIM) | Baseline, Week 26
Change in assessment of QOL using Pediatric Quality of Life Inventory (PedsQL) | Baseline, Week 26
Change in caregiver impression of overall severity of symptoms (behavior and seizure control) using the Caregiver Global Impression of Severity (CareGI-S) | Baseline, Week 4, Week 13, Week 26, Week 52
Change in participant impression of overall severity of symptoms (behavior and seizure control) using the Patient Global Impression of Severity (PGI-S) | Baseline, Week 4, Week 13, Week 26, Week 52
Change in clinician impression of overall severity of symptoms (behavior and seizure control) using the Clinician Global Impression of Severity (CGI-S) | Baseline, Week 4, Week 13, Week 26, Week 52
Retention Rate | Baseline, Week 13, Week 26, Week 52
  Retention rate is the number of participants continuing with CBD-OS treatment over total accrued participants
Number of participants considered treatment responders | Baseline, Week 4, Week 13, Week 26, Week 52
  Treatment responders will be reported as those with a 25%, 50%, 75% and 100% reduction in seizure frequency from baseline
Change in number of seizure-free days | Baseline, Week 4, Week 13, Week 26, Week 52
Number of participants experiencing a worsening, no change, or improvement in seizure frequency | Baseline, Week 4, Week 13, Week 26, Week 52
  Number of participants who experience a change in seizure frequency from baseline defined as:
  1. worsening (>25%)
  2. no change (-25 to + 25%)
  3. improvement (-25% to -50%, ≥-50% to -75%, ≥-75%)
Change in ideation score per the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Week 4, Week 13, Week 26, Week 52
Change in number of suicide attempts per the C-SSRS | Baseline, Week 4, Week 13, Week 26, Week 52
Change in ideation score per the Children's C-SSRS | Baseline, Week 4, Week 13, Week 26, Week 52
Change in number of suicide attempts per the Children's C-SSRS | Baseline, Week 4, Week 13, Week 26, Week 52
Number of participant inpatient hospitalizations due to epilepsy | Up to Week 52
Number of withdrawals due to Treatment Emergent Adverse Events (TEAEs) | Up to Week 52

CONTACTS AND LOCATIONS:
Locations (19):
- United States (12):
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida Health - Department of Neurology, Gainesville, Florida
  - Nicklaus Children's Health, Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minnesota Epilepsy Group, Roseville, Minnesota
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - University of Texas Health Science Center at Houston - Clinical Research Unit, Houston, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Charlottesville, Virginia
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
- The Children's Memorial Health Institute, Warsaw, Poland
- United Kingdom (3):
  - Evelina London Children's Hospital Guys St Thomas' NHS Foundation Trust, the Guy's Hospital, London, England
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No